CLINICAL TRIAL: NCT00764621
Title: Multi-center, Randomized Comparison Study to eVALUatE Outcomes and Resource Needs of Imaging and Treatment Following Primovist-enhanced MRI of the Liver in Comparison to Extracellular Contrast Media (ECCM)-Enhanced MRI and Contrast-enhanced Computed Tomography (CT) in Patients With a History of Colorectal Cancer and Known or Suspected Metachronous Liver Metastases.
Brief Title: Health Economic Evaluation of Primovist-enhanced Liver MRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 91789; 312041 (Other: company internal); 2008-000583-16 (EudraCT Number)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis
Keywords: Gadolinium ethoxybenzyl DTPA; Contrast media; Outcome Assessment (Health Care); Magnetic Resonance Imaging; Tomography, X-Ray Computed; Liver
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Procedure: Primovist MRI
- Arm 2 (Active Comparator)
  Interventions: Procedure: Extracellular contrast media (ECCM) MRI
- Arm 3 (Active Comparator)
  Interventions: Procedure: Contrast-enhanced CT

INTERVENTIONS:
Procedure: Primovist MRI — Contrast-enhanced MRI with an i.v. application of Primovist in the approved dosage
  Arms: Arm 1
Procedure: Extracellular contrast media (ECCM) MRI — Contrast-enhanced MRI with an i.v. application of an approved extracellular contrast medium in the approved dosage
  Arms: Arm 2
Procedure: Contrast-enhanced CT — Contrast-enhanced 3 phase multidetector CT with an i.v. application of an approved iodinated contrast medium in the approved dosage
  Arms: Arm 3

SUMMARY:
Patients with a history of colorectal cancer and known or suspected liver metastases who are scheduled for contrast-enhanced tomographic imaging will be included in this study. After randomization to either Primovist-enhanced MRI, extracellular contrast media (ECCM)-enhanced MRI or contrast-enhanced (CE)-CT outcomes and resource needs of the diagnostic work-up and treatment will be evaluated for each of the three imaging modalities. Main objectives of the study are to assess the proportion of patients for whom further imaging is required to come to a therapy decision and to evaluate the proportion of patients with intraoperatively modified surgical plans after Primovist-enhanced MRI as compared to ECCM-enhanced MRI and CE-CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected metachronous liver metastases secondary to colorectal cancer who are scheduled for further contrast-enhanced tomographic imaging

Exclusion Criteria:

* Patients (men or women) under 18 years of age
* Patients who have received any contrast material within 24 hours before injection of study drug, or who are scheduled to receive any contrast material within 24 hours after injection
* Patients not eligible to contrast media (CM) injection according to product labeling
* Women who are pregnant, lactating or who are of childbearing potential and have not had a negative urine pregnancy test at baseline visit(s)
* Patients scheduled for liver-specific MRI other than Primovist-enhanced MRI, i.e. Multihance-, Teslascan- or SPIO-enhanced MRI
* Patients who are clinically unstable and whose clinical course is unpredictable (e.g. due to previous surgery, acute myocardial infarction)
* Patients with known anaphylactoid or anaphylactic reaction to any contrast media or hypersensitivity to any allergen including drugs
* Patients with a contraindication for MRI or CT.
* Patients with severe renal impairment (eGFR < 30ml/min/1.73m2) or patients on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary variable is the proportion of patients in each of the three treatment groups for whom further imaging is required after initial imaging to come to a therapy decision. | At end of the study (per patient)

SECONDARY OUTCOMES:
Proportion of patients with intra-operatively modified surgical plans based on initial imaging with either Primovist-, ECCM-MRI or CE-CT | After end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (38):
- Austria (3):
  - Vienna, Vienna
  - Graz
  - Vienna
- Germany (9):
  - Karlsruhe, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Greifswald, Mecklenburg-Vorpommern
  - Dortmund, North Rhine-Westphalia
  - Dresden, Saxony
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Italy (6):
  - Candiolo, Torino
  - Ancona
  - Bologna
  - Brescia
  - Chieti
  - Napoli
- Netherlands (3):
  - Amsterdam
  - Leiden
  - Utrecht
- South Korea (5):
  - Seoul, Korea
  - Gyeunggi-do, South Korea
  - Hwasun
  - Jeonbuk
  - Seoul
- Spain (3):
  - Barcelona, Barcelona
  - Santa Cruz de Tenerife, Canary Islands
  - Seville, Sevilla
- Sweden (2):
  - Stockholm
  - Uppsala
- Switzerland (5):
  - Basel, Canton of Basel-City
  - Geneva, Canton of Geneva
  - Lucerne, Canton of Lucerne
  - Sankt Gallen, Canton of St. Gallen
  - Bern
- Thailand (2):
  - Bangkok
  - Songkhla

REFERENCES:
- [Derived] Zech CJ, Korpraphong P, Huppertz A, Denecke T, Kim MJ, Tanomkiat W, Jonas E, Ba-Ssalamah A; VALUE study group. Randomized multicentre trial of gadoxetic acid-enhanced MRI versus conventional MRI or CT in the staging of colorectal cancer liver metastases. Br J Surg. 2014 May;101(6):613-21. doi: 10.1002/bjs.9465. Epub 2014 Mar 20. PMID 24652690
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu